CLINICAL TRIAL: NCT01169402
Title: Safety and Pharmacokinetics of Fluconazole Prophylaxis in Children Supported With Extracorporeal Membrane Oxygenation
Brief Title: Pharmacokinetics/Pharmacodynamics (PK/PD) of Fluconazole in Children on Extracorporeal Membrane Oxygenation (ECMO)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Cohen-Wolkowiez (Other)
Responsible Party: Sponsor-Investigator, Michael Cohen-Wolkowiez, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00022822
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Cardiopulmonary Arrest; Fungal Infection
Keywords: extracorporeal membrane oxygenation; ECMO; extracorporeal life support; fluconazole; diflucan; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Heart Arrest; Mycoses | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluconazole (Experimental)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — 25mg/kg intravenously once weekly while on ECMO
  Other Names: Diflucan

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a form of heart-lung bypass used to support children who suffer heart or lung failure until whatever illness caused that failure can be treated and reversed. While on ECMO, children are at increased risk of infection, including fungal infection. Treatment for fungal infection includes not only antifungal medications but also removal of any large intravenous (IV) lines. Since ECMO requires large IV lines, proper treatment of fungal infections would be difficult if not impossible. The investigators believe that giving prophylactic antifungal medication to all children on ECMO may prevent fungal infections from developing in the first place.

Fluconazole is an antifungal medication that works well against the most common fungal infections and has been shown to be safe in children. Unfortunately, the ECMO machine has the potential to significantly alter the drug levels of medications so the investigators do not know the proper dose of Fluconazole to give children on ECMO. Standard dosing of fluconazole is 12mg per kilogram of body weight given intravenously once daily. Based on preliminary data and modeling from other studies, the investigators think 25mg per kilogram given once weekly will achieve proper drug levels to prevent fungal infections. The investigators have obtained FDA approval to give this dose of fluconazole to children on ECMO who are enrolled in the study. Blood samples will be collected at specific times around the first and second fluconazole doses to describe the PK and drug extraction by the ECMO circuit.

ELIGIBILITY:
Inclusion Criteria:

1. <= 17.5 years at the time of enrollment.
2. Sufficient venous access to permit administration of study medication.
3. Supported with either venoarterial (VA) or venovenous (VV) ECMO.
4. Availability and willingness of the parent/legal guardian to provide written informed consent.

Exclusion Criteria:

1. Subject with a history of anaphylaxis attributed to an azole.
2. Any other concomitant condition, which in the opinion of the investigator would preclude a subject's participation in the study.
3. Previous participation in this study.
4. Subjects who are receiving or who have received cyclosporine, tacrolimus, or azithromycin in the 72 hours prior to first dose of study product require protocol chair notification prior to enrollment.
5. Pregnancy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2013-02-20 (Actual); Study Completion 2013-02-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics/Pharmacodynamics | Quarterly
  Determine proper dosing of fluconazole in children supported with extracorporeal membrane oxygentation

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Watt, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States